CLINICAL TRIAL: NCT05100342
Title: Prospective Validation of a Points Score System Predicting 30-day Survival for Patients With Metastatic Cancer Receiving Palliative Radiation Therapy
Brief Title: Prospective Validation of a Points Score System Predicting 30-day Survival
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Naoyuki G. Saito, M.D., Ph.D., Assistant Professor of Radiation Oncology, Indiana University
Other Study IDs: CTO-IUSCCC-0763
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer
Keywords: palliative radiation; radiation therapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low-risk: Low-risk:score 0-6
  Interventions: Diagnostic Test: Point score prediction tool for 30-day survival
- Intermediate-risk: Intermediate-risk: score 7-13
  Interventions: Diagnostic Test: Point score prediction tool for 30-day survival
- High-risk: High-risk:score 14-20
  Interventions: Diagnostic Test: Point score prediction tool for 30-day survival

INTERVENTIONS:
Diagnostic Test: Point score prediction tool for 30-day survival — This tool requires laboratory data including white blood cell count, neutrophil-lymphocyte ratio, blood urea nitrogen, bilirubin, albumin, lactate dehydrogenase, and red cell distribution, as well as number of attendances to the emergency room in the past 100 days, the site receiving radiation therapy, and the primary cancer type. Each data point correlates with a point value, which are tallied to generate a final score.
  The scores range from 0-20, with 0 giving the highest chance for survival at 30 days and 20 giving the lowest chance for survival at 30 days

SUMMARY:
This is a one-stage single-arm phase II clinical trial designed to prospectively test the survival prediction tool as developed by Lee et al on patients referred to radiation oncology for palliative treatments. Survival prediction score based on objective data including laboratory values, attendance to emergency room, and primary cancer origin will be assigned to each patient at time of enrollment.

DETAILED DESCRIPTION:
This is a one-stage single-arm phase II clinical trial designed to prospectively test the survival prediction tool as developed by Lee et al (section 10.0) on patients referred to radiation oncology for palliative treatments. Survival prediction score based on objective data including laboratory values, visits to emergency room, and primary cancer origin will be assigned to each patient at time of enrollment. The prediction tool assigns a score from 0-20, with 20 indicating the worst survival prognosis; the investigators have designated mortality risk groups as follows: low-risk (score 0-6), intermediate-risk (score 7-13), and high-risk (score 14-20). Patient survival and quality of life will then be monitored at 30-day, 90-day, and 365-day intervals. The study will test the hypothesis that patients with a score of >14 have a less than 20% chance of survival at 30 days.

Primary Objective:

1. To evaluate 30-day survival of patients with a score of >14 (high-risk group)

Secondary Objectives:

1. To evaluate 30-day, 90-day, and 365-day survival of patients in low-risk (score 0-6), and intermediate-risk (score 7-13) groups, and to evaluate 90-day and 365-day survival of patients in high-risk group (score >14)
2. To evaluate patient-reported quality of life at the above intervals using the validated FACIT-Pal-14© questionnaire (Functional Assessment of Chronic Illness Therapy - Palliative Care 14 Item Version)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 at time of consent
2. Ability to provide written informed consent
3. Cancer diagnosis referred to Radiation Oncology for palliative radiation therapy
4. Patients who either choose to not receive radiation therapy or not recommended to receive radiation therapy will remain eligible
5. Those patients who undergo a course of palliative radiation therapy, it is not the requirement of this study to complete that course of treatment. Those who prematurely end their course of treatment will remain eligible Note: Patients who ultimately either choose to not receive radiation or not recommended to receive radiation will remain eligible

Note: Patients who ultimately do not complete prescribed radiation will remain eligible

Exclusion Criteria:

1. Patients who are unable to participate in follow up visits per investigator discretion (virtual/phone follow up is permitted)
2. Patients who are receiving definitive/curative course of radiation therapy
3. Patients who self-report as pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients will be identified and recruited per the recommendation of the consulting radiation oncologist at IUSCCC, IUH Methodist Hospital, Schwarz Cancer Center and IU West hospital.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
30-day survival of patients with a score of >14 (high-risk group) | From baseline to 30 days after enrollment
  The percentage of patients with a score of >14 who are living at 30 days following enrollment

SECONDARY OUTCOMES:
The percentage of patients in each risk group (low, intermediate, and high) who are living at 30 days, 90 days, and 365 days following enrollment | 30 days, 90 days and 365 days after enrollment
  Review of medical records.
Tabulated patient-report quality of life surveys at 30 days, 90 days, and 365 days | Baseline, 30 days, 90 days and 365 days after enrollment
  Using the FACIT-Pal-14© questionnaire (Functional Assessment of Chronic Illness Therapy - Palliative Care 14 Item Version

CONTACTS AND LOCATIONS:
Overall Officials: Naoyuki Saito, MD PhD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - IU Health West, Avon, Indiana
  - IU Health North / Schwarz Cancer Center, Carmel, Indiana
  - Methodist Hospital, Indianapolis, Indiana